CLINICAL TRIAL: NCT02823301
Title: Implementation of VAMOS Program at Health Centers of Florianópolis: Analysis of Different Environments Settings
Brief Title: VAMOS Program at Different Environments of Florianópolis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Aline Mendes Gerage, PhD student, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAMOS 2016
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VAMOS group (Experimental): Active life improving health: all participants that will be assigned to change behavior group will participate of a change behavior program, entitled VAMOS (Active Life Improving Health), for five months. The VAMOS Program is a lifestyle promotion program, that includes physical activity and healthy eating habits. The program is composed by 12 meetings (six weekly meetings and six fortnightly meetings), in group, lasting about 90 min. In each In each weekly meeting, will be discussed guidelines and strategies for physical activities practices in different domains and for adoption of a healthy diet. All aspects and strategies included in the program are based in behavior changes theories.
  Interventions: Behavioral: VAMOS Program
- Control group (No Intervention): Group that will not receive the VAMOS program as intervention.

INTERVENTIONS:
Behavioral: VAMOS Program — Active life improving health: all participants that will be assigned to change behavior group will participate of a change behavior program, entitled VAMOS (Active Life Improving Health), for five months. The VAMOS Program is a lifestyle promotion program, that includes physical activity and healthy eating habits. The program is composed by 12 meetings (six weekly meetings and six fortnightly meetings), in group, lasting about 90 min. In each In each weekly meeting, will be discussed guidelines and strategies for physical activities practices in different domains and for adoption of a healthy diet. All aspects and strategies included in the program are based in behavior changes theories.
  Arms: VAMOS group

SUMMARY:
The main purpose of this study is to evaluate the effectiveness and the maintenance of a behavior change program called VAMOS (Active Life Improving Health) Program on physical activity and healthy eating habits in different environmental contexts of Florianópolis/ SC/ Brazil. This study will be conducted in Health Centers (HC) of Florianópolis/ SC/ Brazil, defined according to environmental and income characteristics. Therefore, initially all geographic areas around the HC will be visited to classify the public places as favorable (with the presence of spaces for the practice of PA) and unfavorable environmental (do not have spaces for physical activity). Thereafter, four HC will be selected: high income + high environmental quality index, high income + low environmental quality index, low income + high environmental quality index, low income + low environmental quality index. In each HC, the volunteers will be randomly assigned into two groups of approximately 25 people: VAMOS group and control group. The participants that will be assigned to the VAMOS group will participate in a behavioral change program aimed at motivating changes in physical activity and eating habits during five months (12 meetings - six weekly meetings and six fortnightly meetings), while the control group will receive one educational lecture regarding lifestyle changes. The meetings of VAMOS Program will be held in the dependences or nearby the HC and will be mediated by the physical education professional previously trained. The Program will be evaluated by the RE-AIM framework: reach, effectiveness, adoption, implementation and maintenance. The effectiveness will be assessed from measurements of physical activity, eating habits, self-efficacy, social support, quality of life, anthropometry, and lipid profile before and after five months of intervention. The implementation will be assessed by identifying the extent to which the program will be conducted as planned. The maintenance will be estimated from revaluations of all outcomes, as measured before and after the intervention, six months and one year after the end of the program.

DETAILED DESCRIPTION:
The main purpose of this study is to evaluate the effectiveness and the maintenance of a behavior change program called VAMOS (Active Life Improving Health) Program on physical activity and healthy eating habits in different environmental contexts of Florianópolis/ SC/ Brazil. This study will be conducted in Health Centers (HC) of Florianópolis/ SC/ Brazil, defined according to environmental and income characteristics. Therefore, initially all geographic areas around the HC will be visited to classify the public places as favorable (with the presence of spaces for the practice of PA) and unfavorable environmental (do not have spaces for physical activity), using the instrument Physical Activity Resource Assessment (PARA). Thereafter, four HC will be selected: high income + high environmental quality index, high income + low environmental quality index, low income + high environmental quality index, low income + low environmental quality index. In each HC, the volunteers will be randomly assigned into two groups of approximately 25 people: VAMOS group and control group, resulting in a total sample of approximately 200 volunteer users. The volunteers will be invited to attend a lecture on healthy lifestyle in date, place and time set, in which a screening will be held in order to trace the profile of the population reached. On this occasion, a questionnaire containing information of sociodemographic data, health status, quality of life, physical activity, eating habits will be answered. They also will be asked to report their individual height and body mass. The participants that will be assigned to the VAMOS group will participate in a behavioral change program aimed at motivating changes in physical activity and eating habits during five months (12 meetings - six weekly meetings and six fortnightly meetings), while the control group will receive one educational lecture regarding lifestyle changes. The meetings of VAMOS Program will be held in the dependences or nearby the HC and will be mediated by the physical education professional previously trained. The Program will be evaluated by the RE-AIM framework: reach, effectiveness, adoption, implementation and maintenance. The effectiveness will be assessed from measurements of physical activity, eating habits, self-efficacy, social support, quality of life, anthropometry, and lipid profile before and after five months of intervention. The implementation will be assessed by identifying the extent to which the program will be conducted as planned. The maintenance will be estimated from revaluations of all outcomes, as measured before and after the intervention, six months and one year after the end of the program. For data analysis, in addition to descriptive statistics, two-way ANOVA for mixed models will be applied for within and between groups comparison, if the premises of this test are met. The level of significance that will be adopted is P<0.05. All analyzes will be done at SPSS statistical package, version 17.0.

ELIGIBILITY:
Inclusion Criteria:

* Must be registered in the public health system;
* Must have been attended on health center at least one time during the last six months;
* Must be classified as " insufficiently active".

Exclusion Criteria:

* Not agree to participated to the study;
* Not agree to sign the written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
change in physical activity | baseline, 5 months, 11 months, 17 months
  Habitual physical activity will be assessed by GT3X or GT3X+ accelerometer (Actigraph - USA) and Actilife 6.10 software will be used to analysis. Each participant will be instructed to use the accelerometer for seven consecutive days, removing it only for sleeping, bathing or performing water activities. The device will be attached to an elastic belt and fixed in the right side of the hip. Data will be collected in a 30 Hz sample frequency and will be analyzed using 60-s epochs. Periods with consecutive values of zero (with 2-min of spike tolerance) for 60 min or longer will be interpreted as "accelerometer not worn" and excluded from the analysis. Physical activity data only will be included if the participant accumulate a minimum of 10 hours/day of recording for at least four days, including one weekend day
change in eating habits | baseline, 5 months, 11 months, 17 months
  Eating habits will be investigated from the score generated by the food frequency questionnaire, using questions from previous studies (Brasil, 2014; Lopes, 2010). The questionnaire will be applied, using a list of foods for which the average frequency of consumption over the last three months is given.

SECONDARY OUTCOMES:
change in body mass | baseline, 5 months, 11 months, 17 months
  The body mass (kg) will be measured according to the recommendations from the International Standards for Anthropometric Assessment (2011)
change in body mass index | baseline, 5 months, 11 months, 17 months
  The body mass index will be calculated with the measurements of body mass and stature that will be measured according to the recommendations from the International Standards for Anthropometric Assessment (2011)
change in waist and hip circumference | baseline, 5 months, 11 months, 17 months
  The waist and hip circumferences (cm) will be measured according to the recommendations from the International Standards for Anthropometric Assessment (2011)
change in self-efficacy for physical activity | baseline, 5 months, 11 months, 17 months
  The self-efficacy for physical activity will be evaluated by a scale proposed by Ammerman et al.(1991).
change in self-efficacy for eating habits | baseline, 5 months, 11 months, 17 months
  The self-efficacy for eating habits will be evaluated by a scale proposed by Ammerman et al.(1991).
change in social-support for physical activity | baseline, 5 months, 11 months, 17 months
  The social support for physical activity will be evaluated by a scale proposed by Reis et al. (2011).
change in social-support for eating habits | baseline, 5 months, 11 months, 17 months
  The social support for eating habits will be evaluated by a scale proposed by Sallis (1987).
change in quality of life | baseline, 5 months, 11 months, 17 months
  The quality of life will be assessed by two general questions from Whoqol BREF.
change in fasting glucose | baseline, 5 months, 11 months, 17 months
  The fasting glucose will be determined by blood sample. Venous blood will be collected in vacuum tubes without anticoagulant following the recommendations for venous blood collection with 12 hours of fasting. These measurements will be performed using diagnostic kits according to the manufacturers instructions respecting the internal quality controls.
change in total cholesterol | baseline, 5 months, 11 months, 17 months
  The total cholesterol will be determined by blood sample. Venous blood will be collected in vacuum tubes without anticoagulant following the recommendations for venous blood collection with 12 hours of fasting. These measurements will be performed using diagnostic kits according to the manufacturers instructions respecting the internal quality controls.
change in HDL-cholesterol | baseline, 5 months, 11 months, 17 months
  The HDL-cholesterol will be determined by blood sample. Venous blood will be collected in vacuum tubes without anticoagulant following the recommendations for venous blood collection with 12 hours of fasting. The concentration of LDL-cholesterol is calculated using the Friedewald formula. These measurements will be performed using diagnostic kits according to the manufacturers instructions respecting the internal quality controls.
change in triglycerides | baseline, 5 months, 11 months, 17 months
  The lipid profile triglycerides will be determined by blood sample. Venous blood will be collected in vacuum tubes without anticoagulant following the recommendations for venous blood collection with 12 hours of fasting. These measurements will be performed using diagnostic kits according to the manufacturers instructions respecting the internal quality controls.

CONTACTS AND LOCATIONS:
Overall Officials: Tania R Benedetti, doctor, Study Director — Federal University of Santa Catarina; Cassiano R Rech, doctor, Study Director — Federal University of Santa Catarina
Locations (1):
- Universidade Federal de Santa Catarina, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Undecided